CLINICAL TRIAL: NCT06964412
Title: A Phase II Randomized Study of the Use of Artificial Intelligence Generated Contours in Ultrasound-based Prostate HDR Brachytherapy
Brief Title: The Use of Artificial Intelligence Generated Contours in Radiation Planning of the Prostate Brachytherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martin King, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Martin King, MD, PhD, Radiation oncologist, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-116
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The experienced clinician will be blinded to the randomization of the contouring method by the new learner. The prostate contour generated by the new learner will then undergo review by the experienced clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MANUALLY GENERATED CONTOURS IN ULTRASOUND-BASED PROSTATE HDR BRACHYTHERAP (No Intervention): Manual prostate contouring by a learner (resident or fellow/new attending) performing prostate HDR brachytherapy.
- AI GENERATED CONTOURS IN ULTRASOUND-BASED PROSTATE HDR BRACHYTHERAPY (Experimental): AI-assisted (U-net algorithm) prostate contouring by a learner (resident or fellow/new attending) performing prostate HDR brachytherapy.
  Interventions: Other: Artificial-intelligence (AI)

INTERVENTIONS:
Other: Artificial-intelligence (AI) — Utilizing the addition of artificial intelligence during prostate contouring.
  Arms: AI GENERATED CONTOURS IN ULTRASOUND-BASED PROSTATE HDR BRACHYTHERAPY

SUMMARY:
This study is investigating how AI can help doctors outline the prostate on an ultrasound image to make a custom radiation plan during a specialized type of radiation treatment for prostate cancer called brachytherapy.

DETAILED DESCRIPTION:
This is a Phase II prospective study evaluating the standard U-net, a deep learning AI algorithm for auto-contouring of the prostate during HDR prostate brachytherapy with the needles in place by new learners. Contouring will be done on TRUS. The study will be conducted with a randomized design. Each patient will be assigned to a new learner and then randomized to manual versus AI-assisted contouring. The randomization will be stratified by new learner type: resident versus fellow/new attending. The hypothesis is that AI-assisted learner contours will have improved Dice coefficients with respect to clinically approved contours compared with manual learner contours. All brachytherapy contours will undergo review by the treating radiation oncologist who is the experienced clinician for clinical approval prior to patient treatment. The experienced clinician will be blinded to the randomization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Deemed suitable candidates for whole gland HDR prostate brachytherapy under general anesthesia as a monotherapy, boost or salvage treatment.

Exclusion Criteria:

* Prior permanent seed LDR brachytherapy implant
* Prior transurethral resection of the prostate (TURP)
* Presence or insertion of a rectal spacer
* Focal HDR brachytherapy treatment i.e. not whole prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinically approved contour vs. Manual and AI assisted contours | 1 day
  Dice coefficient [0: no match, 1: complete match] between the final clinically approved brachytherapy prostate contours versus the manual and AI-assisted contours provided by the new learner.

SECONDARY OUTCOMES:
Contouring time | 1 day
  Contouring time-to-completion needed to generate and edit manual vs AI-assisted contours for a new learner.
Impression of AI or manual contours by new learner | 1 day
  Subjective impressions/perception of AI or manual contours by the new learner based on survey responses.
Impression of AI or manual contours by experienced clinician | 1 day
  Subjective impressions/perception of AI or manual contours by the experienced clinician based on survey responses.
Clinician contours vs. Trus images with and without needles | 1 day
  Dice coefficients of expert clinician contours between TRUS images with implanted needles and TRUS images after removal of bottom needle rows.

CONTACTS AND LOCATIONS:
Overall Officials: Martin King, MD, PHD, Principal Investigator — Dana-Farber Cancer Institute / Brigham Women's Hospital

REFERENCES:
- [Background] Morton G, McGuffin M, Chung HT, Tseng CL, Helou J, Ravi A, Cheung P, Szumacher E, Liu S, Chu W, Zhang L, Mamedov A, Loblaw A. Prostate high dose-rate brachytherapy as monotherapy for low and intermediate risk prostate cancer: Efficacy results from a randomized phase II clinical trial of one fraction of 19 Gy or two fractions of 13.5 Gy. Radiother Oncol. 2020 May;146:90-96. doi: 10.1016/j.radonc.2020.02.009. Epub 2020 Mar 5. PMID 32146259
- [Background] Crook J, Marban M, Batchelar D. HDR Prostate Brachytherapy. Semin Radiat Oncol. 2020 Jan;30(1):49-60. doi: 10.1016/j.semradonc.2019.08.003. PMID 31727300
- [Background] Chen CP, Weinberg V, Shinohara K, Roach M 3rd, Nash M, Gottschalk A, Chang AJ, Hsu IC. Salvage HDR brachytherapy for recurrent prostate cancer after previous definitive radiation therapy: 5-year outcomes. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):324-9. doi: 10.1016/j.ijrobp.2013.01.027. Epub 2013 Mar 6. PMID 23474112
- [Background] Valle LF, Lehrer EJ, Markovic D, Elashoff D, Levin-Epstein R, Karnes RJ, Reiter RE, Rettig M, Calais J, Nickols NG, Dess RT, Spratt DE, Steinberg ML, Nguyen PL, Davis BJ, Zaorsky NG, Kishan AU. A Systematic Review and Meta-analysis of Local Salvage Therapies After Radiotherapy for Prostate Cancer (MASTER). Eur Urol. 2021 Sep;80(3):280-292. doi: 10.1016/j.eururo.2020.11.010. Epub 2020 Dec 11. PMID 33309278
- [Background] Lavoie-Gagnon H, Martin AG, Poulin E, Archambault L, Pilote L, Foster W, Vigneault E, Carignan D, Lacroix F. Advantages of TRUS-based delineation for high-dose-rate prostate brachytherapy planning. J Contemp Brachytherapy. 2022 Feb;14(1):1-6. doi: 10.5114/jcb.2022.113544. Epub 2022 Feb 18. PMID 35233228
- [Background] Podgorsak AR, Venkatesulu BP, Abuhamad M, Harkenrider MM, Solanki AA, Roeske JC, Kang H. Dosimetric and workflow impact of synthetic-MRI use in prostate high-dose-rate brachytherapy. Brachytherapy. 2023 Sep-Oct;22(5):686-696. doi: 10.1016/j.brachy.2023.05.005. Epub 2023 Jun 12. PMID 37316376
- [Background] King MT, Kehayias CE, Chaunzwa T, Rosen DB, Mahal AR, Wallburn TD, Milligan MG, Dyer MA, Nguyen PL, Orio PF, Harris TC, Buzurovic I, Guthier CV. Observer preference of artificial intelligence-generated versus clinical prostate contours for ultrasound-based high dose rate brachytherapy. Med Phys. 2023 Oct;50(10):5935-5943. doi: 10.1002/mp.16716. Epub 2023 Sep 4. PMID 37665729
- [Background] Sullivan GM, Artino AR Jr. Analyzing and interpreting data from likert-type scales. J Grad Med Educ. 2013 Dec;5(4):541-2. doi: 10.4300/JGME-5-4-18. No abstract available. PMID 24454995
- See also: American Cancer Society key statistics for prostate cancer. — https://www.cancer.org/cancer/types/prostate-cancer/about/key-statistics.html
- See also: National Comprehensive Cancer Network. — https://www.nccn.org/professionals/physician_gls/pdf/prostate.pdf

DOCUMENTS (1):
  • Study Protocol (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT06964412/Prot_000.pdf